CLINICAL TRIAL: NCT05210556
Title: Oral Antibiotic Bowel Preparation in Gynecologic Oncology Surgery
Status: Completed | Type: Observational
Sponsor: WellSpan Health (Other)
Responsible Party: Principal Investigator, Eav Lim, Principal Investigator, WellSpan Health
Other Study IDs: 1847220-1
Record Dates: First submitted 2022-01-13; First posted 2022-01-27 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-04

CONDITIONS: Surgical Site Infection; Surgical Complication; Gynecologic Cancer
Keywords: surgical site infection; gynecologic cancer
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- No Antibiotic Bowel Prep: Patients who did not receive a preoperative antibiotic bowel preparation
  Interventions: Other: Diagnosed with Surgical Site Infection
- Antibiotic Bowel Prep: Patients who did receive a preoperative antibiotic bowel preparation

INTERVENTIONS:
Other: Diagnosed with Surgical Site Infection — As an observational study, this notates patients who were diagnosed with a deep organ/space surgical site infection within 30 days of surgery
  Groups: No Antibiotic Bowel Prep

SUMMARY:
The purpose of this study is to investigate whether the use of a preoperative antibiotic bowel regimen is associated with a reduced risk of deep organ/space surgical site infection in gynecologic oncology surgery.

DETAILED DESCRIPTION:
This is a retrospective chart review study. Patients who underwent scheduled intra-abdominal surgery with a WellSpan gynecologic oncologist will be identified and their chart reviewed for demographic data of age, race, BMI, comorbidities, and type of surgery. Those patients who had a deep organ/space surgical site infection within 30 days postoperatively will be identified. The numbers of these infections before and after August 2020, at which time all patients moving forwards were prescribed antibiotic bowel preparation, will then be statistically analyzed and compared to see if the institution of the antibiotic bowel preparation was associated with a reduction in surgical site infection.

ELIGIBILITY:
Inclusion Criteria:

- Underwent scheduled intra-abdominal surgery with a WellSpan gynecologic oncologist

Exclusion Criteria:

* Unscheduled surgery
* Intraoperative consult by a WellSpan gynecologic oncologist

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who had intra-abdominal surgery by a WellSpan gynecologic oncologist from 2019-2021 as identified by review of the surgical schedule.
Sampling Method: Non-Probability Sample
Enrollment: 778 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Surgical Site Infection Rates Associated with Antibiotic Bowel Prep | 2019-2021
  Rate of surgical site infection rate as associated with or without use of antibiotic bowel preparation

CONTACTS AND LOCATIONS:
Locations (1):
- WellSpan, York, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nelson RL, Glenny AM, Song F. Antimicrobial prophylaxis for colorectal surgery. Cochrane Database Syst Rev. 2009 Jan 21;(1):CD001181. doi: 10.1002/14651858.CD001181.pub3. PMID 19160191
- [Background] Morris MS, Graham LA, Chu DI, Cannon JA, Hawn MT. Oral Antibiotic Bowel Preparation Significantly Reduces Surgical Site Infection Rates and Readmission Rates in Elective Colorectal Surgery. Ann Surg. 2015 Jun;261(6):1034-40. doi: 10.1097/SLA.0000000000001125. PMID 25607761
- [Background] Kalogera E, Van Houten HK, Sangaralingham LR, Borah BJ, Dowdy SC. Use of bowel preparation does not reduce postoperative infectious morbidity following minimally invasive or open hysterectomies. Am J Obstet Gynecol. 2020 Aug;223(2):231.e1-231.e12. doi: 10.1016/j.ajog.2020.02.035. Epub 2020 Feb 26. PMID 32112733
- [Background] Nichols RL, Broido P, Condon RE, Gorbach SL, Nyhus LM. Effect of preoperative neomycin-erythromycin intestinal preparation on the incidence of infectious complications following colon surgery. Ann Surg. 1973 Oct;178(4):453-62. doi: 10.1097/00000658-197310000-00008. No abstract available. PMID 4743867